CLINICAL TRIAL: NCT06910995
Title: The Impact of Augmented Reality Location-Based Games on Physical Activity in Middle-Aged and Older Adults.
Brief Title: Augmented Reality Location-Based Games on Physical Activity
Acronym: AR on PA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202412060
Record Dates: First submitted 2025-02-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-01

CONDITIONS: Physical Activity; Quality of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Augmented Reality Location-Based Games (Experimental)
  Interventions: Behavioral: AR location-based game
- Control arm (No Intervention): The control group will maintain their usual routines without any intervention.

INTERVENTIONS:
Behavioral: AR location-based game — This study aims to utilize the AR location-based game Pikmin Bloom to gradually encourage middle-aged and older adults in the community to develop a habit of walking outdoors. A step goal will be set every two weeks to progressively increase daily walking activity. By integrating the AR game with a LINE chatbot for feedback and engagement, this approach aims to motivate older adults, enhance their willingness to go outside, and increase their daily step count.
  Arms: Augmented Reality Location-Based Games

SUMMARY:
This study aims to examine the effects of an augmented reality location-based game intervention on behavioral and psychological factors related to physical activity among middle-aged and older adults. The study adopts a quasi-experimental design, targeting community-dwelling individuals aged 40-59 or 60 and above, who engage in sedentary work patterns exceeding 6 hours daily. Recruitment is scheduled to commence in February 2025 at the Xinyi Health Service Center in Taipei City. Participants will be assigned to either the experimental group or the control group based on enrollment timing. A minimum of 41 participants will be recruited, divided into two experimental groups and two control groups. The experimental group will participate in an augmented reality location-based game featuring different step count goals every two weeks, daily step count reporting, and goal achievement encouragement. The control group will maintain their usual routines without any intervention. The intervention will last for 8 weeks. Research instruments will include a basic demographic questionnaire, the short-form Taiwan Physical Activity Questionnaire, the Exercise Self-Efficacy Scale, the Exercise Motivation and Barriers Scale, blood pressure measurements, and the Quality of Life Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Meet one of the following conditions: middle-aged to senior citizens aged 40 to 59 years old or senior citizens aged 60 years old or older who work more than 6 hours a day in a sedentary lifestyle
2. Able to walk independently without the use of aids.
3. Have a smart phone with an application (Pikmin Bloom) that can be installed and can access the Internet and GPS.

Exclusion Criteria:

1. Patients who have been diagnosed by a doctor as suffering from dementia, mental illness or major diseases.
2. Those who are unable to do intense exercise as mentioned in the medical advice.
3. Those who cannot go out for long time, such as family caregivers.
4. Those who have regular exercise habits: average daily steps over 5,000 steps or 30 minutes of leisure-type physical activity more than 3 times a week.
5. Those who will not use the AR adaptive game (Pikmin Bloom) at the end of the 2-day test period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire short-form | Baseline, through study completion, an average of 12 weeks
  It consists of 7 items that ask about physical activity over the last 7 days. These items cover vigorous activities, moderate activities, walking, and sitting (MET-minute/week)
Exercise Self-Efficacy Scale | Baseline, through study completion, an average of 12 weeks
  Participants achieved a response if they scored an exercise self-efficacy score between 1 and 10.
The Exercise Motivation and Barriers Scale | Baseline, through study completion, an average of 12 weeks
  It typically includes a series of statements related to exercise benefits and barriers. Participants rate their agreement with each statement on a Likert scale (5 strongly agree to 1 strongly disagree)
WHO Quality of Life Scale. | Baseline, through study completion, an average of 12 weeks
  A shorter version with 26 questions. The scale evaluates various aspects of life, including physical health, psychological state, social relationships, and environmental factors, scored between 1 and 5.

SECONDARY OUTCOMES:
Blood pressure | Baseline, through study completion, an average of 12 weeks
  Electronic blood pressure monitor
Body composition | Baseline, through study completion, an average of 12 weeks
  Tanita Body composition monitors

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan